CLINICAL TRIAL: NCT06985563
Title: Exacerbation of Erythema Following PDT in Patients With Probable Capillary Malformation-Arteriovenous Malformation Syndrome: Retrospective Analysis of Ultrasound and Clinical Characteristics.
Status: Completed | Type: Observational
Sponsor: Second Affiliated Hospital of Xi'an Jiaotong University (Other)
Responsible Party: Principal Investigator, Weihui Zeng, Professor, Second Affiliated Hospital of Xi'an Jiaotong University
Other Study IDs: 2024213
Record Dates: First submitted 2025-05-14; First posted 2025-05-22 (Actual); Last update posted 2025-05-22 (Actual); Status verified 2025-05

CONDITIONS: Probable Capillary Malformation-Arteriovenous Malformation Syndrome
Keywords: exacerbation of erythema following PDT; probable CM-AVM syndrome; Ultrasound; retrospective study

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Exacerbation of erythema following PDT group: Patients experiencing exacerbation of clinical symptoms, such as darker coloration than before treatment, following at least one Hemoporfin-PDT session were recruited.
  Interventions: Combination Product: HMME-PDT; Device: Ultrasound examinations

INTERVENTIONS:
Combination Product: HMME-PDT — Prior to treatment, patients or their guardians provided written informed consent. Then patients were then prepared for the procedure by fully exposing the treatment area and shielding the surrounding normal skin with a black cloth. Hemoporfin (Shanghai Fudan-Zhangjiang Bio-Pharmaceutical) was administrated intravenously at a dosage of 5.0 mg/kg. Subsequently, patients underwent light radiation at 532 nm (Wuhan Yage Optic and Electronic Technique, Wuhan, China) for 18 to 25 minutes, with a power density randing form 75 to 110 mW/cm2.
Device: Ultrasound examinations — Ultrasound examinations were performed using three types of devices: a Paragon XHD equipped with a L38-22 probe operating at a frequency of 20-30 MHz (Kolo Medical Co., Ltd, Suzhou, China), a DUB Skin Scanner with a 22 MHz probe (Taberna Pro Medicum, German), or a Mindray Resona 7 featuring an L14-5WU linear probe set to a frequency range of 11-12 MHz frequency (Mindray Bio-Medical Electronics Co., Ltd, Shenzhen, China).

SUMMARY:
This study aims to reduce the misdiagnosis rate of PWSs and improve the diagnosis of CM-AVM using ultrasound. Furthermore, we seek to provide more evidence-based recommendations for the treatment of patients with probable CM-AVM syndrome, particularly those presenting with erythema.

DETAILED DESCRIPTION:
Background: Exacerbation of erythema following photodynamic therapy (PDT) in patients with probable capillary malformation-arteriovenous malformation (CM-AVM) syndrome, may be attributed to misdiagnosis as port-wine stains (PWSs).

Objective: To identify the ultrasound features of patients with exacerbation of erythema following PDT for a definite diagnosis.

Methods: A retrospective single-center study was conducted on PWS patients with exacerbation of erythema following PDT. The clinical and ultrasonic features were reviewed and analysed. One low-frequency and two high-frequency ultrasound (HFUS) devices were used to examine the lesions and the contralateral normal skin.

Results: The clinical characteristics of 16 patients were consistent with those of high-flow vascular stains (HFVS). Ultrasound findings revealed skin and hypodermis thickening, increased blood flow signals with an arteriovenous malformation (AVM) waveform and deeper, larger blood vessels in the dermis and hypodermis of pink macules (PMs) compared to normal skin. In the absence of genetic diagnosis, PWS patients with exacerbation of erythema following PDT were diagnosed as having probable CM-AVM syndrome.

Limitations: Retrospective single-center design and small sample size. Conclusion: Patients with PWSs are advised to undergo low-frequency ultrasound examinations to avoid misdiagnosis. HFUS can serve as a complementary method to promptly identify underlying AVMs beneath the PMs. We do not recommend PDT treatment for patients with probable CM-AVM syndrome.

ELIGIBILITY:
Inclusion Criteria:

* Patients who were greater than or equal to 1 year old at the time of their first HMME-PDT treatment.

  * Patients who experiencing exacerbation of clinical symptoms, such as darker coloration than before treatment.

    * Patients who have undergone one or more HMME-PDT treatments. ④ Patients with complete basic information and treatment-related information.

Min Age: 1 Year | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients experiencing exacerbation of clinical symptoms, such as darker coloration than before treatment, following at least one Hemoporfin-PDT session were recruited between 2017 and 2023 at the Department of Dermatology, Second Affiliated Hospital of Xi'an Jiaotong University.
Sampling Method: Non-Probability Sample
Enrollment: 16 (Actual)
Dates: Start 2024-03-01 (Actual); Primary Completion 2024-06-01 (Actual); Study Completion 2024-06-01 (Actual)

PRIMARY OUTCOMES:
ultrasound characteristics | The efficacy evaluation will be conducted 3 months after the completion of the 1st HMME-PDT treatment.
  After cleaning and disinfecting the mesured area, the probe, coated with 1-2 millimeters of coupling agent, was positioned vertically on the skin surface. Measurements of skin thickness, density, vessel diameter, and depth were obtained for both the lesions and the contralateral normal skin. The color Doppler (CD) mode of high-frequency ultrasound was employed to assess local blood perfusion in both lesions and normal skin, while the pulsed-wave (PW) Doppler mode was used to detect the blood flow spectrum. The average of three measurements at the same site was calculated.

CONTACTS AND LOCATIONS:
Overall Officials: Weihui Zeng, Study Chair — Second Affiliated Hospital of Xi'an Jiaotong University
Locations (1):
- The Second Affiliated Hospital of Xi'an Jiaotong University, Xi'an, Shaanxi, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Rodriguez Bandera AI, Feito Rodriguez M, Chiloeches Fernandez C, Stewart N, Valdivielso-Ramos M. Role of colour-Doppler high-frequency ultrasonography in capillary malformation-arteriovenous malformation syndrome: a case series. Australas J Dermatol. 2020 Nov;61(4):349-352. doi: 10.1111/ajd.13311. Epub 2020 May 3. PMID 32363619
- [Background] Cen Q, Sun Y, Zeng X, Liu Y, Liu F, Chen H, Lin X, Cai R. Unilateral and segmental distribution of facial erythema: is it a real port-wine stain? Hereditas. 2020 Jul 7;157(1):27. doi: 10.1186/s41065-020-00143-z. PMID 32635943
- [Background] Valdivielso-Ramos M, Torrelo A, Martin-Santiago A, Hernandez-Nunez A, Azana JM, Campos M, Berenguer B, Garnacho G, Moreno R, Colmenero I. Histopathological hallmarks of cutaneous lesions of capillary malformation-arteriovenous malformation syndrome. J Eur Acad Dermatol Venereol. 2020 Oct;34(10):2428-2435. doi: 10.1111/jdv.16326. Epub 2020 May 19. PMID 32124491
- [Background] Liu J, Zhou J, Hu D, Cui L, Li Y, Ye D, Wu T, Mi B, Geng S, Zeng W. Retrospective analysis of Hemoporfin-mediated photodynamic therapy in the treatment of naive port-wine stains. Photodiagnosis Photodyn Ther. 2022 Sep;39:103003. doi: 10.1016/j.pdpdt.2022.103003. Epub 2022 Jul 13. PMID 35840007